CLINICAL TRIAL: NCT00258024
Title: Control of Pregnancy Associated Malaria With Intermittent Preventive Treatment Through Community Involvement in Rural Ghana
Brief Title: Control of Pregnancy Associated Malaria With Intermittent Preventive Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ghana5.2.malaria
Record Dates: First submitted 2005-11-23; First posted 2005-11-24 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Anaemia; Malaria
Keywords: IPT-SP, pregnancy, malaria,Ghana
MeSH Terms: conditions — Anemia; Malaria

INTERVENTIONS:
Drug: IPT-sulphadoxinepyrimethamine

SUMMARY:
Malaria is one of the major causes of illness and mortality in Sub-Saharan Africa. In Ghana, malaria is the most important cause of morbidity and accounts for about 40% of outpatient contacts. Chemoprophylaxis and insecticide-impregnated bed nets are used for malaria control in pregnancy.Chloroquine is administered within the ANC package at health facilities in Ghana. However, many pregnant women in rural,low-income communities do not report for ANC or report late thereby increasing their risk of morbidity and mortality. Reasons for this include inaccessibility and high cost. As the gap between urban and rural health care and socioeconomic circumstances increase, malaria control remains the major challenge of the health sector. A facility-based intervention alone is not sufficient to have a significant or sustained impact on malaria control in pregnancy. Alternative strategies are needed for the delivery of malaria interventions to pregnant women in rural areas in Ghana. The overall objective of this study is to develop alternative strategies for community involvement for delivery of malaria interventions to pregnant women in rural Ghana. The project will be conducted in the Afigya Sekyere district in the Ashanti Region of Ghana. Interviews and focus group discussions will be conducted with pregnant women and community members focusing on local knowledge on control of malaria in pregnancy and factors influencing utilization of antenatal services. Women in their first and second pregnancies who are permanently resident in the study area will be included in the study using IPT with sulphadoxine-pyrimethamine (SP). The study population will be randomized to:Group 1 will receive clinic-supervised IPT-SP and daily folate/iron supplementation and Group 2 will access IPT-SP with daily folate/iron supplementation from trained traditional birth attendants (TBA). Midwives and TBAs will be trained in preparing thick blood smears and placenta biopsies for parasitological examination. Parasitaemia and Hb will be measured at entry and at delivery and fever episodes during pregnancy will be recorded. Study participants will be followed for adverse reactions within a week after drug administration. The effectiveness of community-based IPT for the control of malaria in pregnancy will be determined. The endpoints of the study will be birth weight, maternal anaemia, fever episodes and prevalence of peripheral and placental parasitaemia in the groups.

DETAILED DESCRIPTION:
General Objective To evaluate an alternative strategy of community involvement in the control of pregnancy associated malaria and anaemia in an area of intense malaria transmission in Ghana.

Specific Objectives To explore local knowledge and health-care practices of control of malaria in pregnancy and determine factors influencing utilization of antenatal services by pregnant women.

To determine the prevalence of malaria and anaemia in pregnancy in the Afigya Sekyere district To determine the effect of intermittent preventive treatment on pregnancy outcome in primigravidae and secundigravidae To evaluate the effectiveness of a health facility and a community-based malaria intervention in first and second pregnancies

Methodology Study area and population The study will be conducted in the Afigya Sekyere district of the Ashanti Region of Ghana. The district lies within the forest belt where malaria prevalence is highest (AHMED, 1989). Mean temperature is 270C with annual rainfall between 1500 and 2000mm. The major rainfall season is between March-July and the minor in September - November. There is little seasonal variation in malaria parasite transmission and rates are just slightly higher after the rains. Most of the inhabitants are peasant farmers.The district is divided into six sub districts with 91 communities.It has 15 health facilities (2 hospitals, 6 health centres, 2 clinics and 5 maternity homes). The district has about 42 trained (TTBAs) and a number of untrained TBAs who conduct almost 30% of deliveries in the district (DHA, 2002).Considering the inadequate number of health professionals coupled with their exodus to developed countries, the capabilities of TBAs can be enhanced and used in control of malaria in pregnancy.

Study Design Pre-intervention phase A baseline Survey on birth weights will be carried out to determine the mean birth weight and birth weight distribution in the study area

Qualitative data collection Focus group discussions (FGDs) and interviews will be conducted at health facilities and in communities to explore local knowledge on control of malaria in pregnancy and social, cultural and economic factors influencing utilization of antenatal and delivery services by pregnant women. This will involve pregnant women of all parities, village health committee members, TBAs and opinion leaders.

Cross-sectional Survey (determination of prevalence of parasitaemia and anaemia) A cross-sectional survey will be conducted to determine the prevalence of parasitaemia and anaemia among pregnant women in the district. Pregnant women will be randomly selected from health institutions and six communities. The sample at the health facility will be women used for the exit interview. Twenty percent of pregnant women from six communities will be used. Their blood samples will be taken for parasitaemia rate and density and their haemoglobin levels will be measured using a Haemocue.

Intervention phase

This phase will involve Community-based and Health Facility-based administration of single-dose SP (1500/75mg) to pregnant women and assess its effect on the following outcome:

Birth weight Anaemia Parasitaemia Fever episodes

Sample Size:420 women of first and second pregnancy. Selection of field sites and training of staff Using random sampling, 20 TTBAs will be selected from communities without health facilities. Six health facilities will also be purposively selected as field sites. Two field supervisors (FS) will be employed to help with the study. They will be trained in data collection, interviewing, monitoring drug administration, preparing blood smears, checking haemoglobin and weighing of babies.

A one-week training session will be organized for the selected TTBAs. They will be trained in:

Drug storage and administration Interviewing Recognizing imminent complications in pregnancy Taking placenta biopsy and making thick blood smears Weighing of babies Record keeping

A one-day meeting will also be held with the heads of the health institutions and all the midwives in the district to brief them on the study and solicit their support. Midwives from the 10 selected health facilities will later be trained in:

Taking placental biopsy and making thick blood smears Haemoglobin measurements Interviewing Record keeping

3) Enrolment of Study Participants

The inclusion criteria for this phase are women who are:

primigravidae or secundigravidae have Hb >7g/dl (Those with Hb below 7g/dl will be treated and later enrolled) permanently resident in the district no reaction to sulpha drugs no multiple pregnancy no chronic diseases

Midwives and TTBAs will recruit women at ANCs and in communities, confirm non-palpable pregnancies by testing their urine and interview them for reaction to sulpha drugs. The researcher, laboratory technician and FS will visit field sites, gather background information from the women and check their gestation, haemoglobin and parasitaemia levels to obtain baseline data for each woman. Eligible women who give their consent by signing or thumb-printing a consent form will be enrolled into the study and given identification cards. They will be advised to present this card to the midwives anytime they visit an antenatal clinic so that no antimalarial will be given them as prophylaxis.

3) Drug administration Group 1 - Health Facility Intervention (HFI) Midwife supervised IPT with daily iron and folate supplementation. Women in this group will receive single-dose treatment with sulphadoxine-pyrimethamine (1500/75mg) twice in the second trimester at least one month apart and once in the third trimester when they visit the antenatal clinic. This will begin from 16 weeks gestation. They will also receive daily iron and folate supplementation. They will be informed to immediately report to the health facility with any adverse effects they might experience.

Group 2- Community-Based Intervention (CBI) TTBA supervised IPT with daily iron and folate supplementation. Women in this category will receive sulphadoxine-pyrimethamine (1500/75mg) and daily iron and folate supplementation from 16 weeks gestation. Two doses of this anti-malarial will be taken during the second trimester at least one month apart and a third dose early in the third trimester under the supervision of the TTBA. The women will be instructed to immediately report any adverse reactions to the health facility and the TTBA, which will be recorded. The TTBAs will be encouraged to promptly refer women with imminent complications to health facilities for appropriate treatment.

4) Laboratory investigations The midwives, TTBAs and FS will have regular supply of slides, slide boxes, gloves, cotton wool and methanol to prepare and store blood smears and placenta biopsies. All blood samples from midwives and TTBAs will be collected weekly by FS and transported to Kwame Nkrumah University of Science and Technology for processing and microscopic examination by a laboratory technician. Haemoglobin and parasitaemia values will be compared for the groups. Ten (10%) percent of the slides will be read at Komfo Anokye Teaching Hospital in Kumasi for quality control.

5) Delivery Scales will be provided for TTBAs and health facilities without reliable scales to weigh babies and record their birth weight. There will be regular monitoring visits by the researcher and FS to ensure accurate recording of birth weights. Providers will be supplied with forms and notebooks for record keeping. The birth weights in the two groups will be compared.

6) Referrals A follow-up will be made for records on women who develop pregnancy-related complications and are referred to health facilities outside the district.

Ethical considerations

1. Ethical clearance for the study will be sought from the following:

   * Committee on Human Research Publications and Ethics of the School of Medical Sciences, KNUST.
   * Ashanti Regional Health Administration (ARHA)
   * Afigya Sekyere DHMT.
   * Danish Central Ethical Committee
2. Eligible women will be asked to give their consent before participation and confidentiality of information gathered will be ensured.
3. Women who develop pregnancy-related complications would be referred to health facilities that are equipped to handle such cases and the cost of their treatment will be borne by the project. All health facility in-charges will be informed about this.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida
* Secundigravida
* Permanent resident
* Hemoglobin (Hb) > 7 g/dl

Exclusion Criteria:

* Hb < 7 g/dl
* Allergy to sulpha
* Multiple pregnancy
* Chronic diseases

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 420 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Birth weight
anaemia
parasitaemia
fever episodes

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Bam, reg. nurse, Principal Investigator — Dept. Community Health, School of Health Sciences, Kumasi University
Locations (1):
- Afiya Sekyere district, Kumasi, Ashanti Region, Ghana

REFERENCES:
- See also: Related Info — http://www.dblnet.dk